CLINICAL TRIAL: NCT02706041
Title: Damage Control Laparotomy: A Randomized Controlled Trial
Brief Title: Damage Control Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, John Andrew Harvin, MD, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-GEN-16-0104; UL1TR000371 (NIH); KL2TR000370 (NIH)
Record Dates: First submitted 2016-02-27; First posted 2016-03-11 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Other Injury of Other Intra-abdominal Organs, Initial Encounter
Keywords: Exploratory Lap (Ex Lap); Damage Control Laparotomy (DCL); Definitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Definitive closure laparotomy (Active Comparator): Subjects randomized to the definitive closure laparotomy arm will have the incision closed at the end of the exploratory laparotomy.
  Interventions: Procedure: Definitive Closure Laparotomy
- Damage control laparotomy (Other): Subjects randomized to the damage control laparotomy arm will have the incision left open at the end of the exploratory laparotomy. The trauma team will evaluate the patient's clinical course to determine when the incision can be closed.
  Interventions: Procedure: Damage Control Laparotomy

INTERVENTIONS:
Procedure: Definitive Closure Laparotomy — Subjects randomized to the definitive closure laparotomy arm will have the incision closed at the end of the exploratory laparotomy.
  Arms: Definitive closure laparotomy
Procedure: Damage Control Laparotomy — Subjects randomized to the damage control laparotomy arm will have the incision left open at the end of the exploratory laparotomy. The trauma team will evaluate the patient's clinical course to determine when the incision can be closed.
  Arms: Damage control laparotomy

SUMMARY:
Randomized study to compare outcomes of patients undergoing damage control laparotomies versus definitive closure for which there is surgeon equipoise to randomize.

DETAILED DESCRIPTION:
Single center, prospective, randomized study involving seriously injure patients requiring an emergent laparotomy within 90 minutes of arrival to the emergency department. There are situations in which the patient is unable to be closed at the end of the emergent laparotomy (identified as damage control) and there are situations in which the injury has been treated and the incision can be closed (definitive). There are also situations where it is not clear if the patient should be kept open or closed and the result of the surgery varies based on the surgeon performing the case.

The eligible subjects for this study will be randomized toward the end of the emergent laparotomy procedure on a 1:1 basis and will be followed throughout the hospitalization for complications. Patients will also be contacted at 6 month to complete a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Emergent laparotomy
* Patient has injuries for which surgeon has equipoise to perform a Definitive (DEF) or Damage Control Laparotomy (DCL)
* Age ≥16 years (age cut-off for admission to adult trauma service at Memorial Hermann Hospital-Texas Medical Center)

Exclusion Criteria:

* Indication for DCL for which there is no surgeon equipoise:

  * Need for gauze packing of liver or retroperitoneum for hemorrhage control
  * Immediate need to go to Interventional Radiology for hemorrhage control
  * Concern for Abdominal Compartment Syndrome - defined as physically unable to re-approximate fascia or >10mmHg change in peak airway pressure during fascial closure
  * Hemodynamic instability - defined as persistent hypotension, ongoing transfusion requirement, or continuous vasopressor use
* Indication for DEF for which there is no surgeon equipoise:

  * Negative and non-therapeutic laparotomies
  * Isolated cystorrhaphy
* Prisoners
* Known pregnancy
* Patients with burns > 20% of total body surface area
* Patient/legally authorized representative opted out of exception from informed consent (opt out bracelet)
* Currently enrolled in another interventional study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Harvin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvin JA, Podbielski J, Vincent LE, Fox EE, Moore LJ, Cotton BA, Wade CE, Holcomb JB. Damage control laparotomy trial: design, rationale and implementation of a randomized controlled trial. Trauma Surg Acute Care Open. 2017 Apr 13;2(1):e000083. doi: 10.1136/tsaco-2017-000083. eCollection 2017. PMID 29766087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Started | 18 | 21
Received Allocated Intervention | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 40] | 29 [24 to 48] | 30 [24 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 14 | 17 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 7 | 3 | 10
  Race/Ethnicity: Hispanic | 5 | 7 | 12
  Race/Ethnicity: White | 6 | 1 | 7
  Race/Ethnicity: Other | 0 | 10 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 21 | 39
Mechanism of Injury [Count of Participants; unit: Participants]
  Blunt | 10 | 12 | 22
  Penetrating | 8 | 9 | 17
Area of Injury [Count of Participants; unit: Participants]
  Liver | 10 | 10 | 20
  Spleen | 10 | 11 | 21
  Kidney | 6 | 7 | 13
  Small Bowel | 8 | 9 | 17
  Large Bowel | 6 | 7 | 13
  Pancreas | 3 | 7 | 10
  Stomach | 3 | 5 | 8
  Major Venous Injury | 0 | 1 | 1
  Major Arterial Injury | 1 | 0 | 1
  Femur | 4 | 4 | 8
  Pelvis | 7 | 8 | 15
  Traumatic Brain Injury | 5 | 6 | 11
Grade of Liver Injury [Median (Inter-Quartile Range); unit: units on a scale] — Grade ranges from 1 to 5, with a higher grade indicating worse injury
  units on a scale | 3 [2 to 3] | 2 [1 to 3] | 3 [2 to 3]
Grade of Spleen Injury [Median (Inter-Quartile Range); unit: units on a scale] — Grade ranges from 1 to 5, with a higher grade indicating worse injury
  units on a scale | 3 [1 to 3] | 4 [2 to 5] | 3 [2 to 4]
Grade of Kidney Injury [Median (Inter-Quartile Range); unit: units on a scale] — Grade ranges from 1 to 5, with a higher grade indicating worse injury
  units on a scale | 2 [1 to 4] | 4 [3 to 5] | 4 [2 to 4]
Score on Abbreviated Injury Scale (AIS) - Head [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 0 [0 to 4] | 1 [0 to 3] | 0 [0 to 4]
Score on Abbreviated Injury Scale (AIS) - Chest [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 3 [1 to 3] | 3 [0 to 3] | 3 [0 to 3]
Score on Abbreviated Injury Scale (AIS) - Abdomen [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 4 [3 to 4] | 3 [3 to 4] | 3 [3 to 4]
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: score on a scale] — The Injury Severity Score (ISS) assesses the combined effects of injuries in multiple anatomical locations and ranges from from 1 to 75, with 75 being the most severe.
  score on a scale | 29 [22 to 41] | 34 [20 to 43] | 33 [20 to 43]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died or Had Major Abdominal Complication (MAC)
Description: Major abdominal complication (MAC) is defined as development of an organ/space surgical site infection, enteric suture line failure, fascial dehiscence, or unplanned return to operating room (OR).
Time Frame: 30 days
Population: Analysis is intention to treat, so all who were assigned to the intervention are analyzed, regardless of whether they received the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 18 | 21
Participants
  Death or Major abdominal complication (MAC) | 6 | 12
  Major abdominal complication (MAC) | 6 | 8
  Death | 0 | 7

2. Secondary Outcome: Number of Participants With Non-abdominal Morbidities
Description: Non-abdominal Morbidities include Acute Kidney Failure, Deep Vein Thrombosis, Pulmonary Embolism, Pneumonia, and Urinary Tract Infection.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 18 | 21
Participants
  Number of Participants with Acute Kidney Failure | 3 | 7
  Number of Participants with Deep Vein Thrombosis | 0 | 2
  Number of Participants with Pulmonary Embolism | 1 | 1
  Number of Participants with Pneumonia | 6 | 8
  Number of Participants with Urinary Tract Infection | 3 | 1

3. Secondary Outcome: Number of Hospital-free Days
Description: Number of days patient was not in hospital within the 30 day time frame.
Time Frame: 30 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 18 | 21
days | 13 [0 to 19] | 0 [0 to 11]

4. Secondary Outcome: Number of ICU-free Days
Description: Number of days patient not in the ICU during the 30 day time frame
Time Frame: 30 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 18 | 21
days | 24 [0 to 25] | 12 [0 to 24]

5. Secondary Outcome: Number of Ventilator-free Days
Description: Number of days patient not on ventilator in the 30 day time frame
Time Frame: 30 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 18 | 21
days | 27 [3 to 28] | 22 [0 to 27]

6. Secondary Outcome: Hospital Costs
Time Frame: 30 days
Reporting Status: Not Posted

7. Secondary Outcome: Patient-centered Outcomes Assessed Using the Standard Gamble
Description: Participants are asked to choose between two hypothetical outcomes: 1 - the sure outcome, that is, remaining in a state of ill health for a period of time; or 2 - the gamble, that is, choosing a medical intervention which has a certain probability of either restoring them to perfect health or killing them. The Standard Gamble identifies the probability (of the intervention delivering perfect health) at which the two alternatives (1 and 2) seem equally attractive. Scores range from 0% to 100%, with a score of 100% indicating that a choices 1 and 2 are equally attractive only when there is a 100% probability that the intervention will deliver perfect health, and a score of 0% indicating that choices 1 and and 2 are equally attractive even when there is a 0% probability that the intervention will deliver perfect health.
Time Frame: at discharge from hospital (about 20 days after intervention)
Population: These data were not collected from 6 in the Damage control laparotomy arm and 10 in the Definitive closure laparotomy arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 12 | 11
score on a scale | 2.2 (5.0) | 0.4 (1.0)

8. Secondary Outcome: Patient-centered Outcomes Assessed Using the Standard Gamble
Description: as for outcome 7
Time Frame: 6 months after discharge from hospital
Population: These data were not collected from 6 in the Damage control laparotomy arm and 9 in the Definitive closure laparotomy arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 12 | 12
score on a scale | 9.5 (16.8) | 1.7 (12.7)

9. Secondary Outcome: Patient-centered Outcomes Assessed Using the 5-level European Quality of Life Scale-5D (EuroQol-5D-5L)
Description: The EuroQol-5D-5L assesses health-related quality of life. Total score ranges from 0 to 100, with 0 indicating the worst health imaginable and 100 indicating the best health imaginable.
Time Frame: at discharge from hospital (about 20 days after intervention)
Population: These data were not collected from 2 in the Damage control laparotomy arm and 9 in the Definitive closure laparotomy arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 16 | 12
score on a scale | 19 (33) | 25 (33)

10. Secondary Outcome: Patient-centered Outcomes Assessed Using the 5-level European Quality of Life Scale-5D (EuroQol-5D-5L)
Description: as for outcome 9
Time Frame: 6 months after discharge from hospital
Population: These data were not collected from 5 in the Damage control laparotomy arm and 9 in the Definitive closure laparotomy arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 13 | 12
score on a scale | 55 (36) | 49 (40)

11. Secondary Outcome: Patient-centered Outcomes Assessed Using the Post-Traumatic Stress Disorder Check List - Civilian (PCL-C)
Description: The PCL-C assesses Post-Traumatic Stress Disorder (PTSD) symptoms. Total score ranges from 17-85. A score of 17-29 shows little to no PTSD symptoms. A score of 28-29 indicates some PTSD symptoms. A score of 30-44 indicates moderate to moderately high severity of PTSD symptoms. A score of 45-85 indicates high severity of PTSD symptoms.
Time Frame: at discharge from hospital (about 20 days after intervention)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 13 | 12
score on a scale | 35 (14) | 32 (15)

12. Secondary Outcome: Patient-centered Outcomes Assessed Using the Post-Traumatic Stress Disorder Check List - Civilian (PCL-C)
Description: as for outcome 11
Time Frame: 6 months after discharge from hospital
Population: These data were not collected from 7 in the Damage control laparotomy arm and 8 in the Definitive closure laparotomy arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
Number analyzed (Participants) | 11 | 13
score on a scale | 39 (16) | 31 (11)

ADVERSE EVENTS:
Time Frame: From time of hospital admission to time of discharge from hospital (about 8 to 31 days)
Arm/Group | Damage Control Laparotomy | Definitive Closure Laparotomy
All-Cause Mortality (participants affected / at risk) | 0/18 | 7/21
Serious Adverse Events (participants affected / at risk) | 11/18 | 16/21
Other Adverse Events (participants affected / at risk) | 6/18 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Damage Control Laparotomy (N=18) | Definitive Closure Laparotomy (N=21)
Death (General disorders) | 0 (0) | 7 (7)
Organ/space surgical site infection (Infections and infestations) | 5 (5) | 8 (8)
Fascial dehiscence (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Reopening after closure (Surgical and medical procedures) | 2 (2) | 6 (6)
Sepsis (Immune system disorders) | 9 (9) | 11 (11)
Acute renal failure (Renal and urinary disorders) | 3 (3) | 7 (7)
Multi-organ failure (General disorders) | 4 (4) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Damage Control Laparotomy (N=18) | Definitive Closure Laparotomy (N=21)
Ileus (Gastrointestinal disorders) | 6 (6) | 7 (7)
Pulmonary embolus (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Superficial surgical site infection (Infections and infestations) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
Small sample size; failure to accrue targeted sample size of 56; inability to blind; imbalance of baseline characteristics in randomized arms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02706041/Prot_SAP_000.pdf